CLINICAL TRIAL: NCT04219423
Title: Feasibility and Preliminary Efficacy of Multi-modal Physical Therapy on Physical Performance and Health -Related Quality of Life in Hispanic Older Adults With Moderate Knee Osteoarthritis: a Pilot Study
Brief Title: Feasibility of Multi-modal Physical Therapy in Latino Older Adults With Moderate Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Amy Gladin, Senior Physical Therapist, Kaiser Permanente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN-16-2740_04
Record Dates: First submitted 2019-12-31; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Arthritis Knee
Keywords: Hispanic American; Physical Therapy; Pilot study; Latino

STUDY DESIGN:
Intervention Model Description: This is a small, prospective pre/post evaluation study to determine feasibility for a larger clinical trial. Participants will be recruited from an electronic medical record search and from primary care providers. Recruitment, retention and adherence will be determined. Baseline and post intervention outcomes on physical function and quality of life will be determined for preliminary estimates of change.
Masking Description: Small study staff precludes blinding of assessors and instructors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multimodal physical therapy (Experimental): The multimodal intervention is 75 minutes in duration and meets two days per week for two weeks, then once per week for six weeks, followed by weekly phone calls to determine adherence to home-exercise program (HEP) for four weeks. The total duration of the intervention is twelve weeks. The intervention will be led in a group format with a ratio of one physical therapist to two participants and groups never exceeding 4 participants. All verbal and written communications in the intervention will be conducted in Spanish. The multimodal intervention consists of progressive lower extremity strengthening training targeting the quadriceps and gluteal groups in both legs, progressive stationary bicycle exercise, self-management training and education, manual therapy and home exercise program (HEP) instruction. Participants are asked to do their strengthening exercises at least three days per week for the 12-week study duration including sessions in the clinic
  Interventions: Behavioral: Multimodal physical therapy

INTERVENTIONS:
Behavioral: Multimodal physical therapy — see description in arm/group description

SUMMARY:
This is a small, pilot, pre/post evaluation study enrolling older Hispanic American adults with moderate knee arthritis to evaluate the feasibility of recruitment, retention and adherence after a multimodal 12-week, physical therapy intervention. The secondary aim is to evaluate preliminary estimates of change on physical performance and health related quality of life after the intervention.

DETAILED DESCRIPTION:
Background: Hispanic Americans (HAs) experience more pain and mobility deficits associated with knee osteoarthritis (OA) compared to non-Hispanic whites (NHWs) and seek total knee arthroplasties at a reduced rate, thus conservative treatments are needed. Prevalence of knee OA among the older HA population is rising dramatically. There is moderate evidence that lower extremity strengthening, manual therapy and self-management training improve pain and physical performance in people with knee OA and little evidence in the HA population. We conducted a pilot prospective trial implementing a multimodal high intensity targeted strength training, manual therapy and self-management education intervention to evaluate feasibility of recruitment, retention and adherence and preliminary estimates of change on physical performance and health related quality of life (HrQOL) in HAs with moderate knee OA. If this trial is feasible and shows promise for efficacy, it may warrant further testing as a primary treatment for knee OA.

Methods: Spanish speaking older adults will be recruited from Kaiser Permanente San Francisco through a medical record search. Participants will attended 10 physical thearpy clinic visits over 8 weeks, followed by 4 weekly phone calls to assess adherence to exercise via 1-week verbal recall. Participants will be instructed to exercise 3 days per week for the study duration combining both clinic and home exercise participation. The intervention is led in Spanish and will include progressive open and closed-chain quadriceps and gluteal strengthening, progressive cycling training with short power intervals, manual therapy and self-management training.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate knee osteoarthritis Defined as Kellgren-Lawrence radiographic level 2 or 3
2. People who speak Spanish as a primary language
3. Age 50 or greater
4. pass a Phone screening: Reports problems with physical performance due to knee: Answers yes to 'Are you now limited in any way in any of your usual activities because of arthritis or joint?' Reports pain in their knee: Answers 'yes' to have you had pain in your knee in last 30 days? Be able to walk inside home without a cane, be able to walk ¼ of a block without a cane and be able to go up a flight of stairs without assistance from another

Exclusion Criteria:

1. Psychiatric or behavioral comorbidity preventing participation in a group exercise program
2. History of lower extremity joint arthroplasty
3. Morbid obesity defined as body mass index of 40 or greater
4. Presence of inflammatory arthritic condition
5. Neurologic involvement impacting functional mobility

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-10 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled in the study | 12 weeks
  Number of participants enrolled in to the study to determine ability to recruit for the study.
Percentage of enrolled participants at end of study | 12 weeks
  Number of participants who complete the study divided by the number who enroll in the study to determine retention.
Average number of completed exercise session per-week for the study duration. | 12 weeks
  Number of clinic session attendance plus the number of self-reported participation in home exercise divided by the study goal of exercising 3 days per week for the 12 week study duration (36 exercise sessions total) yielding a percentage to determine adherence to the exercise intervention.

SECONDARY OUTCOMES:
Change in Five-times Sit to Stand (5TSTS) from baseline to after the intervention. | 12 weeks
  5TSTS is a physical performance measure and is the time in seconds it takes for participants to stand up and sit down from a chair 5 times as fast as possible. Shorter duration in seconds indicates improved physical performance.
Change in Six-minute Walk Test (6MWT) from baseline to after the intervention. | 12 weeks
  6MWT is a physical performance measure and is the distance in meters participants are able to walk for 6 minutes at self-selected speed. Shorter distance in meters indicates improved physical performance.
Change in Timed Up and Go (TUG) from baseline to after the intervention. | 12 weeks
  Timed up and go (TUG) is a physical performance measure and is measured in seconds, the time it takes for participants to rise from a chair, walk 10-meters at their 'normal' speed and return to a sitting position. Shorter duration in seconds indicates improved physical performance.
Change in absolute isometric bilateral quadriceps strength physical performance measure from baseline to after the intervention. | 12 weeks
  Absolute isometric quadriceps strength is a physical performance measure and is measured in pounds and normalized to body weight and expressed as a percentage. Quadriceps strength is measured in a sitting position, with participants knee bent to 90 degrees. The examiner stabilizes a hand-held dynamometer on a table leg with a gait-belt strap and aligns the hand held dynamometer 1 inch proximal to the distal fibula on the anterior aspect of the tibia underneath the gait belt. Participants are given 2 to 3 practice sessions on 1 minute rests. Participants are given verbal encouragement to push as hard as they can for 2 trials on 1 minute rests and the average peak force in pounds is recorded. Increased peak force normalized to body-weight percentage indicates improvement in quadriceps strength.
Change the Western Ontario McMaster University Osteoarthritis Index (WOMAC) questionnaire score from baseline to after the intervention. | 12 weeks
  The Western Ontario McMaster University Osteoarthritis Index (WOMAC) is a self-administered questionnaire that measures health-related quality of life in people with lower extremity dysfunction. The WOMAC has 24 questions in total and aggregates constructs of pain (5 questions), stiffness (2 questions) and physical function (17 questions) yielding a maximum score of 96 points. Each question is scored 0 to 4 where 0 indicates 'none' and 4 indicates 'extreme'. Higher scores indicate worse pain, stiffness and physical function. Each construct can be scored separately to represent a single construct.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Gladin, Principal Investigator — Kaiser Permanente

IPD SHARING:
Plan to Share IPD: Yes
Investigators may have a PDF copy of the study protocol upon request or a de-identified data set upon request.
Supporting Information: Study Protocol, CSR
Time Frame: December 20 2019 to December 31 2020.
Access Criteria: Investigators or clinicians can have access to the study intervention protocol or a de-identified data set on outcome measures.